CLINICAL TRIAL: NCT05892172
Title: Characteristics of Arrhythmia and Heart Rate Variability in Patients With Heart Failure and Sleep Disordered Breathing
Brief Title: Heart Failure and Sleep Disordered Breathing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yihui Kong (Other)
Responsible Party: Sponsor-Investigator, Yihui Kong, Professor, First Affiliated Hospital of Harbin Medical University
Organization: First Affiliated Hospital of Harbin Medical University (Other)
Other Study IDs: 2021020707
Record Dates: First submitted 2023-05-18; First posted 2023-06-07 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure
Keywords: sleep disordered breathing; arrhythmia; heart rate variability
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFrEF group: HFrEF was defined as Left ventricular ejection fraction ≤40%
- HFmrEF group: HFmrEF was defined as Left ventricular ejection fraction 41%~49%
- HFpEF group: HFpEF was defined as Left ventricular ejection fraction ≥50%

SUMMARY:
The purpose of this study is to analyze and summarize the characteristics of arrhythmia and heart rate variability of Chinese patients with three different types of heart failure combined with sleep disordered breathing based on the clinical data, to provide new diagnosis and treatment ideas for domestic patients, and then to improve the prognosis of patients betterly.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. The diagnosis of heart failure conforms to the criteria of the Chinese Guidelines for the Diagnosis and Treatment of Heart Failure .
3. Echocardiography, dynamic electrocardiogram and polysomnography monitoring should be improved during the period of hospitalization.
4. Patients with sleep apnea have not received standard treatment.

Exclusion Criteria:

1. Patients undergoing cardiac surgery in the past 6 weeks.
2. Patients with acute decompensated heart failure or heart failure requiring oxygen therapy.
3. All patients with sleep apnea who receive standard treatment.
4. Patients who use pacemakers or implantable cardioverter defibrillators.
5. The patient did not complete the echocardiography, dynamic electrocardiogram, and polysomnography monitoring during hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heart failure patients hospitalized in the Department of Cardiology of the First Affiliated Hospital of Harbin Medical University
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-28 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
heart failure and sleep apnea | 24 hours
  analyze and summarize the characteristics of arrhythmia and heart rate variability of Chinese patients with three different types of heart failure combined with sleep-disordered breathing based on the clinical data. Collection of clinical data: general clinical data, physical signs, post-admission inspection indicators, and treatment conditions of patients collected from the electronic medical record system. Echocardiographic data mainly included ejection fraction, left atrial anterior-posterior diameter, and interventricular septum thickness, which were in millimeters; electrocardiogram examination mainly included Diagnosis type of arrhythmia by dynamic, the overall standard deviation of normal sinus R-R interval (SDNN), the average standard deviation of normal sinus R-R interval throughout the recording period (SDANN), which were in a millisecond, etc; The type and severity of sleep-disordered breathing and Apnea hypopnea index were obtained by polysomnography.

CONTACTS AND LOCATIONS:
Locations (1):
- Yihui Kong, Harbin, Heilongjiang, China